CLINICAL TRIAL: NCT02979938
Title: Understanding Excretion and Infectivity of Zika Virus in Semen During and After Infection
Status: Completed | Type: Observational
Sponsor: Trinidad and Tobago IVF and Fertility Centre (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: ZIKAFERTI
Record Dates: First submitted 2016-11-17; First posted 2016-12-02 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Zika Virus
MeSH Terms: conditions — Zika Virus Infection | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Semen analysis and semen PCR for Zika virus — Every two weeks subjects provide a semen sample which is analysed and then frozen for RT-PCR and viral load. Semen sample testing for the presence of ZIKV (Institute of Tropical Medicine, Belgium) will be performed using both a ZIKV-specific, in-house duplex real-time RT-PCR, targeting a 102bp and 121bp sequence of the NS5 gene and the RealStar® Zika Virus RT-PCR Kit (Altona). Quantitative viral load RNA measurements will be expressed utilizing threshold cycle values because a standardized viral load reference method is not available. To test for infectivity of ZIKV in semen, ZIKV isolation will be attempted in semen samples with a high viral ZIKV load (i.e. positive ZIKV PCR result and Ct-values below 30) by inoculation in Vero cells.

SUMMARY:
In this prospective observational study the investigators will report on 20 male subjects with proven WHO-classification Zika infection. These subjects will be followed up for a maximum of 12 months to observe the presence, viral load and infectivity of Zika virus (ZIKV) in semen over time.

DETAILED DESCRIPTION:
In this prospective observational study the investigators will report on 20 male subjects with proven WHO-classification Zika infection. These subjects will be followed up for a maximum of 12 months to observe the presence, viral load and infectivity of Zika virus (ZIKV) in semen over time.

Knowledge of the possible presence, infectivity and persistence of ZIKV in semen will provide evidence-based data for

1. estimating of the risk of sexual transmission of ZIKV in the general population
2. antenatal guidelines for the prevention of sexual transmission of ZIKV to the fetus
3. advising couples on the length of time that pregnancy should be avoided in women wishing to conceive after their partner's ZIKV infection
4. strategies to prevent transmission of ZIKV infection through assisted reproductive treatment (ART)
5. advice on gamete cryopreservation
6. optimising investigations for diagnosis of ZIKV in males.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18-50 years
* ZIKV symptoms within the preceding thirty days
* Confirmed ZIKV infection (WHO criteria)
* Able to ejaculate to produce a semen sample

Exclusion Criteria:

• Current urological malignancy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 25 men aged 18-50 years with ZIKV symptoms within the preceding thirty days & confirmed ZIKV infection (WHO criteria). The study setting is a private fertility clinic in Trinidad and Tobago - a country with a current ZIKV epidemic.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the presence (with RT-PCR) of ZIKV in semen | 6 months

SECONDARY OUTCOMES:
Measurement of the viral load (with ct values) of ZIKV in semen | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Minto-Bain, MB ChB MRCOG, Principal Investigator — Trinidad & Tobago IVF & Fertility Centre
Locations (1):
- Trinidad and Tobago IVF & Fertility Centre, Maraval, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No